CLINICAL TRIAL: NCT02522910
Title: An Open-label Phase Ib/II Study of BAY 1000394 (Roniciclib) in Combination With Docetaxel in Second- or Third-line Treatment of Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0274
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: NSCLC (Non-Small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — roniciclib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roniciclib with Docetaxel (Experimental)
  Interventions: Drug: BAY 1000394 (Roniciclib) in combination with docetaxel

INTERVENTIONS:
Drug: BAY 1000394 (Roniciclib) in combination with docetaxel — The study (Phase Ib part and Phase II part) will be conducted as a single center study. This study part will be conducted in an open-label, non-randomized, Phase I conventional 3+3 dose-escalating design to define the safety, tolerability, pharmacokinetics, and MTD of BAY 1000394 (Roniciclib) given in a 3 days on / 4 days off schedule in combination with docetaxel in subjects with second- or third-line NSCLC.

SUMMARY:
This study part will be conducted in an open-label, non-randomized, Phase I conventional 3+3 dose-escalating design to define the safety, tolerability, pharmacokinetics, and MTD of BAY 1000394 (Roniciclib) given in a 3 days on / 4 days off schedule in combination with docetaxel in subjects with second- or third-line NSCLC.

DETAILED DESCRIPTION:
This study part will be conducted in an open-label, non-randomized, Phase I conventional 3+3 dose-escalating design to define the safety, tolerability, pharmacokinetics, and MTD of BAY 1000394 (Roniciclib) given in a 3 days on / 4 days off schedule in combination with docetaxel in subjects with second- or third-line NSCLC.

The number of subjects treated in the dose-escalation part depends on the number of dose- escalation or de-escalation steps needed to determine the MTD of BAY 1000394 (Roniciclib) in combination with docetaxel in this subject population.

Subjects treated at the recommended phase II dose level within the Phase Ib part of the study will be included in the response evaluation of the Phase II part.

ELIGIBILITY:
Inclusion Criteria:

Screening must be performed within 14 days prior to the first dose of study drug. Subjects are eligible for inclusion in this study if all of the following criteria are met:

* Histologically or cytologically confirmed stage IIIB or IV NSCLC Patients who received prior 1 or 2 lines of systemic anticancer therapy. For EGFR mutated or ALK rearranged patients, EGFR TKI or ALK inhibitor is also considered a line of systemic therapy
* Documented progressive disease after platinum-containing doublet chemotherapy (Platinum-containing chemotherapy given as an neoadjuvant/adjuvant chemotherapy, or definitive concurrent chemoradiotherapy within 6 months can be considered as one line of chemotherapy)
* For patients who showed non-progressive disease with 1st line platinum-doublet chemotherapy, continuation maintenance therapy is not considered a line of therapy, whereas switch maintenance therapy is considered another line of therapy.
* EGFR mutated or ALK rearranged patients can be eligible after one line of EGFR TKI or ALK inhibitor and platinum-doublet chemotherapy.
* Any prior systemic anticancer therapy must have been completed at least 3 weeks prior to initiation of study medication. Palliative radiation, whole brain radiotherapy (WBRT), or gamma knife surgery (GKS) for brain metastases must have been completed at least 2 weeks prior to initiation of study medication. Major or minor surgery must have been completed at least 4 or 2 weeks prior to initiation of study medication, respectively. Majority or minority of surgery can be decided at the investigator's discretion. Any acute toxicity must have recovered to Grade ≤ 1 (except alopecia).
* Male or female subjects aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements to be conducted within 14 days prior to the first dose of study drug:
* At least one measurable lesion based on RECIST 1.1
* Availability of tumor tissue for molecular analysis is not mandatory (presence of archival tissue or re-biopsy for acquisition of tumor tissue is strongly recommended)

Exclusion Criteria:

Subjects are to be excluded from the study if they display any of the following criteria:

* Prior radiotherapy (local palliative radiotherapy is permitted but must have occurred ≥2 weeks and subject must have no Grade 3 or 4 toxicities prior to first dose of study treatment; palliative is defined as not intended to cure but to relieve symptoms and reduce suffering)
* Eligibility for local therapy (surgery or radiotherapy)
* Previous treatment with any CDK inhibitors or docetaxel
* Current or ongoing administration of anticoagulation or antiplatelet therapy. However, use of low-dose aspirin (≤100 mg/day) and/or low-dose heparin is permitted unless it is being used for conditions other than cancer
* Known hypersensitivity to any of the study treatments or excipients of the preparations or any agent given in association with this study
* Previous deep vein thrombosis (within the last 6 months), arterial thrombotic events (including strokes), or pulmonary embolism
* History of cardiac disease: Congestive heart failure New York Heart Association (NYHA) Class III or IV angina (within past 6 months prior to study entry), myocardial infarction, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Active clinically serious infections of NCI-CTCAE v4.0 >Grade 2
* Known human immunodeficiency virus infection, active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
* Seizure disorder requiring therapy (such as steroids or anti-epileptics)
* Symptomatic metastatic brain or meningeal tumors, including those of the spinal cord, and including cases of neoplastic meningitis (also known as symptomatic carcinomatous meningitis or leptomeningeal carcinomatosis). However, after WBRT or GKS for symptomatic brain or leptomeningeal metastases, if subjects are stable for 2 weeks without steroid and the dosage of anti-convulsant is stable for 2 weeks, they are eligible. Asymptomatic central nervous system metastases are eligible if the subject has no abnormal findings on neurologic examination and is not receiving corticosteroid therapy to control symptoms.
* History of organ allograft
* Evidence or history of bleeding disorder, ie any hemorrhage / bleeding event of NCI-CTCAE v4.0 >Grade 2 within 4 weeks prior to the first dose of study treatment
* Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management)
* Serious, non-healing wound, ulcer, or bone fracture (bone fractures due to bone metastases are acceptable)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 months after the study enrollment
  Determination of the maximum tolerated dose (MTD) of BAY 1000394 (Roniciclib) in combination with docetaxel.
Dose-Limiting Toxicities (DLT) | 4 months after the study enrollment
  Determination of the dose-limiting toxicities (DLT) of BAY 1000394 (Roniciclib) in combination with docetaxel.
Progression-Free Survival (PFS) | 4 months
  Evaluation of the progression-free survival (PFS) at 4 months by RECIST 1.1 criteria.